CLINICAL TRIAL: NCT00745342
Title: Optimizing Adherence and Glycemia in Youth With New IDDM
Brief Title: Optimizing Adherence and Glycemia in Youth With New Insulin-dependent Diabetes Mellitus (IDDM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lori Laffel, Chief, Pediatric, Adolescent, & Young Adult Section; Investigator, Genetics & Epidemiology Section, Joslin Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 92-23; R01DK046887 (NIH)
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes; glycemic control; family conflict; quality of life; parental involvement
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teamwork Group (Experimental): Families randomized to the Teamwork Group received the behavioral family teamwork intervention.
  Interventions: Behavioral: Family Teamwork Intervention
- Standard Care (No Intervention): Families in the Standard Care group received standard diabetes care and equal attention from study staff between visits to schedule appointments and encourage regular diabetes follow-up care.

INTERVENTIONS:
Behavioral: Family Teamwork Intervention — Families in the teamwork group received quarterly psychoeducational interventions at regular clinic visits, focusing on promoting family teamwork and reducing diabetes-specific family conflict and diabetes burnout.
  Arms: Teamwork Group

SUMMARY:
This 2-year randomized, controlled trial examined the impact of a clinic-based, family teamwork intervention on glycemic control in youth with recently diagnosed type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 17 years old
* Duration of type 1 diabetes between 2 months and 6 years
* Residence in New England or New York
* At least 1 outpatient visit in the past year

Exclusion Criteria:

* Major co-morbid psychiatric or medical illness in youth
* Diagnosis of an active major psychiatric disorder in either parent
* Diagnosis of a life-threatening medical illness in either parent

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 1999-03; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Glycemic control, assessed by hemoglobin A1c | 2 years
  Change in A1c from baseline to 2 years, measured every 3 months

SECONDARY OUTCOMES:
Youth quality of life, measured using the youth PedsQL survey and the parent-proxy PedsQL survey | 2 years
  Measured at baseline, 1 year, and 2 years
Diabetes-specific family conflict, measured using the Diabetes Family Conflict survey (youth and parent versions) | 2 years
  Measured at baseline, 1 year, and 2 years
Parent involvement in diabetes management tasks, measured using the Diabetes Family Responsibility Questionnaire (youth and parent versions) | 2 years
  Measured at baseline, 1 year, and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lori MB Laffel, MD, MPH, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Anderson BJ, Vangsness L, Connell A, Butler D, Goebel-Fabbri A, Laffel LM. Family conflict, adherence, and glycaemic control in youth with short duration Type 1 diabetes. Diabet Med. 2002 Aug;19(8):635-42. doi: 10.1046/j.1464-5491.2002.00752.x. PMID 12147143
- [Result] Laffel LM, Vangsness L, Connell A, Goebel-Fabbri A, Butler D, Anderson BJ. Impact of ambulatory, family-focused teamwork intervention on glycemic control in youth with type 1 diabetes. J Pediatr. 2003 Apr;142(4):409-16. doi: 10.1067/mpd.2003.138. PMID 12712059
- [Result] Laffel LM, Connell A, Vangsness L, Goebel-Fabbri A, Mansfield A, Anderson BJ. General quality of life in youth with type 1 diabetes: relationship to patient management and diabetes-specific family conflict. Diabetes Care. 2003 Nov;26(11):3067-73. doi: 10.2337/diacare.26.11.3067. PMID 14578241